CLINICAL TRIAL: NCT05706415
Title: Enhanced Deep Learning Model for Diagnosis of Pancreatic Solid Lesions Through Multimodal Clinical Images
Brief Title: AI Assisted the Diagnosis of Pancreatic Solid Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Changhai Hospital (Other)
Collaborators: The Third People's Hospital of Chengdu (Other); Ruijin Hospital (Other); Sun Yat-sen University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-AI and MDT
Record Dates: First submitted 2023-01-21; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: AI Assist in the Diagnosis of Pancreatic Solid Lesions

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with solid lesions of pancreas
  Interventions: Diagnostic Test: Clinicians will review the suggestions of a hypothetical AI

INTERVENTIONS:
Diagnostic Test: Clinicians will review the suggestions of a hypothetical AI — There is no intervention. Clinicians will review the suggestions of a hypothetical AI

SUMMARY:
Solid lesions of the pancreas mainly include tumor and non tumor lesions. More than 90% of pancreatic tumor lesions are pancreatic cancer, which is characterized by high mortality and poor prognosis and requires surgical treatment; Non-tumor lesions of the pancreas are mainly inflammatory lesions, which usually do not require surgical treatment, but can be treated with drugs. The common ones are chronic pancreatitis and autoimmune pancreatitis, with a good prognosis. Clinically, the differential diagnosis between them is very difficult. Multi-disciplinary diagnosis and treatment of MDT makes our understanding of pancreatic diseases increasingly rich and in-depth. From disease diagnosis to preoperative evaluation and curative effect evaluation, non-invasive imaging involves almost every link under MDT mode. In view of this, improving the differential diagnosis of pancreatic solid space-occupying lesions on imaging will be more conducive to the diagnosis and treatment under MDT mode, so new technologies such as artificial intelligence should be considered. Our goal is to develop a clinically applicable artificial intelligence system, which uses multiple modes to simulate the routine clinical workflow and assist in the diagnosis of benign and malignant pancreatic solid space-occupying lesions.

DETAILED DESCRIPTION:
The diagnosis of solid pancreatic lesions is challenging, MDT is a very effective method, but it has a certain misdiagnosis rate. This is a multi-center, prospective and observational clinical study. Our goal is to develop a clinically applicable artificial intelligence system. On the one hand, our artificial intelligence based on clinical data+CT imaging images can assist MDT doctors to diagnose the nature of pancreatic space-occupying lesions and reduce misdiagnosis; On the other hand, if a patient needs EUS-FNA puncture, the multimodal artificial intelligence system based on clinical data+CT+EUS developed by us can help MDT doctors understand the nature of pancreatic space-occupying lesions and reduce the probability of misdiagnosis or secondary puncture.

ELIGIBILITY:
Inclusion Criteria:

* pancreatic solid mass in CT and EUS

Exclusion Criteria:

* insufficient imaging quality of CT or EUS
* endoscopic ultrasound non accessible lesions

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who had pancreatic solid mass will be enrolled in our study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-21 (Estimated); Primary Completion 2023-02-21 (Estimated); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Researchers use artificial intelligence (AI) support system to assist in diagnosis of pancreatic solid space-occupying lesions | 2 months
  A multi-layer screening deep convolution network based on deep convolution network was developed to observe its accuracy, sensitivity and specificity in assisting MDT doctors to identify benign and malignant pancreatic space-occupying lesions.

CONTACTS AND LOCATIONS:
Locations (1):
- CT and EUS, Shanghai, Shanghai Municipality, China